CLINICAL TRIAL: NCT00911417
Title: The Jetstream G2 System Post-Market Peripheral Vascular IVUS Study
Brief Title: A Study to Collect Intravascular Ultrasound Images Before and After Treatment With the Jetstream System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pathway Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC09030
Record Dates: First submitted 2009-05-19; First posted 2009-06-01 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: peripheral arterial disease; peripheral vascular disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pathway Jetstream Atherectomy System — The Pathway Jetstream System is a commercially available rotating, aspirating, expandable catheter for active removal of plaque and blood clots in peripheral arteries of the lower limbs.

SUMMARY:
The Jetstream System is a commercially available rotating, aspirating, expandable catheter designed to remove atherosclerotic plaque and blood clots in the lower limbs. The purpose of this study is to use intravascular ultrasound (IVUS) during the interventional procedure to measure the amount of plaque and blood clots removed by the Jetstream System.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years of age.
* The documented peripheral vascular disease is/are located in a superficial femoral, popliteal or tibial peroneal trunk arteries in the lower limb.
* The patient is an acceptable candidate for percutaneous intervention using the Jetstream G2 System in accordance with its labeled indications and instructions for use.
* The patient has been informed about the nature of the study and has provided informed consent.

Exclusion Criteria:

* Patient has no distal runoff.
* Interventional treatment is intended for in-stent restenosis at the peripheral vascular site.
* Patient is pregnant or nursing a child.
* Intended interventional treatment includes planned laser, brachytherapy or atherectomy procedure other than the Jetstream G2 System.
* Patient has clinically significant abnormal ECG or blood test results or any other factor that would put the patient at increased risk if participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plaque Morphology | up to 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tom Davis, MD, Principal Investigator — St. John's Hospital and Medical Center
Locations (5):
- United States (5):
  - Arizona Heart Institute, Phoenix, Arizona
  - St. Luke's Hospital, Phoenix, Arizona
  - St. John's Hospital, Springfield, Illinois
  - St. John Hospital & Medical Ctr., Detroit, Michigan
  - Mount Sinai Medical Center, New York, New York